CLINICAL TRIAL: NCT06844877
Title: Italian NCL Registry: a Registry for NCL as an Integration Tool for Future Therapeutic Strategies
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Filippo Maria Santorelli, Director of Molecular Medicine, IRCCS Fondazione Stella Maris
Other Study IDs: Italian NCL Registry
Record Dates: First submitted 2025-02-10; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Neuronal Ceroid Lipofuscinosis
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood, urine, skin biopsy, muscle biopsy, cerebrospinal fluid (all samples are optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal is to create a solid and harmonious disease registry of patient affected by neuronal ceroid lipofuscinosis (NCLs) that facilitates the collection and management of patients' data over time encouraging the research and the development of future clinical trials. In-depth clinical phenotyping will develop significant clinical outcome measures that can be used in clinical trials and will allow the phenotypic complexity of the disease to be captured with the use of validated clinical scales, biomarkers and so-called patient reported outcomes (PROs).

DETAILED DESCRIPTION:
The registry will involve three recruiting clinical centres (IRCCS Fondazione Stella Maris in Pisa, Ospedale pediatrico Bambin Gesù in Roma e IRCCS Istituto Neurologico Carlo Besta in Milano). Participants will be assessed annually at one of the three participating clinical sites. For each patient, at least one follow-up visit will be scheduled at an interval of 12 months in order to monitor and compare the longitudinal progression of NCLs in similar groups (for example based on phenotype, age at onset, or genotype). At each visit all enrolled subjects will carry out a clinical-instrumental evaluation as per clinical practice, including: anamnestic collection, general and neurological objective examination; administration of illness scales (e.g. the Hamburg scale, UBDRS) and questionnaires about psychiatric symptoms, sleep disorders and quality of life. Any biological samples will be collected as tissues, blood or urine and stored in the laboratories or bio-repositories of the individual centers and also reported in the electronic clinical report form (CRF) of NCL Registry. The results of further diagnostic tests carried out such as Optical coherence tomography (OCT), brain magnetic resonance imaging (MRI) or neurophysiology performed during diagnostic practice or clinical follow up will also be collected. Any further clinical scales/evaluation questionnaires to be administered will be selected according to clinical need based on the neurological characteristics and genotype of each participant. All data relating to further instrumental and/or neurophysiological investigations carried out by the patient for clinical needs will also be collected.

The data collected during the aforementioned clinical-instrumental-laboratory evaluations will be entered into the Italian NCL registry in pseudonymized form.

ELIGIBILITY:
Inclusion Criteria:

* genetically confirmed diagnosis of neuronal ceroid lipofuscinosis
* participants/parents/legal guardians will have to give informed consent for enrollment in the registry and privacy data management

Exclusion Criteria:

* subjects affected by other forms of neurodegenerative diseases.
* lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects affected by NCLs with a genetic or ultrastructural characterization
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-07-19 (Estimated); Study Completion 2027-07-19 (Estimated)

PRIMARY OUTCOMES:
Establishment of the NCL Italian Registry to systematically document the clinical presentation and natural history of patients affected by NCLs | 12 months
  We will record information related to NCL natural history in 10 patients

CONTACTS AND LOCATIONS:
Overall Officials: Filippo M Santorelli, Dr., Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- IRCCS Fondazione Stella Maris, Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data collected during the clinical-instrumental-laboratory evaluations will be entered into the Italian NCL Registry in pseudonymized form. Each patient will be identified by a progressive code of the electronic CRF together with a unique alphanumeric identification code (automatically generated). This identification code will be used by the Center in place of the relevant name in each communication of the linked data. The Recruiting Center will be the only and exclusive entity able to associate the identification code with the personal data. The data collected in the Italian NCL Registry will be stored on RedCap in pseudonymized form.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: january 2027
Access Criteria: Collaborative research centers working on NCL